CLINICAL TRIAL: NCT05648344
Title: WW Improving Nutrition Study: A Randomized Controlled Trial
Acronym: WINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Southern University (Other)
Collaborators: WW International Inc (Industry); Indiana University (Other)
Responsible Party: Principal Investigator, Ana Palacios, Assistant Professor, Georgia Southern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H23120
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Overweight and Obesity
Keywords: behavioral weight management; digital health; diet quality
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to WW app for 6 months (Experimental): Participants will be randomized to access the WW application for 6 months
  Interventions: Behavioral: WW
- Control (Placebo Comparator): Participants will be randomized to receive emails with information available from myplate.gov
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: WW — WW assigns foods to a point value calculated through a proprietary algorithm that accounts for the food's caloric value, saturated and unsaturated fat, sugar, fiber, and protein. Members are encouraged to track their food and beverage intake, with the goal of staying within their personal points targets assigned based in an individual's sex, age height, weight, goals, and activity. The program also has "Zero Point Foods" (list of healthy foods with no point value) and can be eaten freely. In addition to the personal points, participants will be asked to attend WW coach-led virtual workshops conducted over Zoom, engage with peer- support, and WW-trained behavior change experts via 24/7 chat.
  Arms: Access to WW app for 6 months
Behavioral: Control — Usual care with information from myplate.gov
  Arms: Control

SUMMARY:
The main objective of this study is to determine whether a behavior change weight management and wellness program (WW) delivered via an app for 6-months will be effective in improving diet quality in U.S. adult participants, relative to a control group through a randomized controlled trial.

DETAILED DESCRIPTION:
The WW Unlimited Workshops and Digital Program is an evidence-based behavioral weight management program that guides members toward personal weight and wellness goals through a personalized curriculum, complemented with behavioral weekly goals to drive healthy habits. The program includes foods that can be eaten in moderation without the need to tracking, as well as a points system that rates foods. In addition, members have access to food, activity, water, sleep, and weight trackers, meal planning tools, recipes, guided meditations and workouts, peer support, and access to online workshops and WW-trained behavior change coach.

To compare the 6-month changes in diet quality (HEI-2015 total score), in adult participants enrolled in a commercial weight-loss program (WW) vs. control, a total of 376 adults will be recruited via social media and other online platforms in the contiguous 48 States of the US. Participants will be randomly assigned to access the WW app, or a control, and will be followed-up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported desire to lose weight
* English proficiency
* Ages: 18 - 70 years old
* BMI between 27-45 kg/m2
* Owns a smartphone with a camera
* Wi-Fi connectivity at home
* Willing to follow recommendations required by study protocol
* Willing to actively participate in a behavioral weight loss program for 6 months and to attend virtual workshop meetings
* Willing to include demographic information (e.g., ethnicity, income, and education)
* US residence (48 contiguous States)
* Must be able to receive in the mail a weight scale.

Exclusion Criteria:

* Pregnant, lactating, or plans to become pregnant during study period
* Self-reported bipolar disorder, substance abuse, psychosis, bulimia.
* Meets criteria for severe depression on the Patient Health Questionnaire-8 (PHQ-8) (score of >20)
* All other mental health, including other eating disorders will be assessed using a self-report question on the initial screening survey.
* Had bariatric surgery or plans to have any surgery during the study
* Unable or not willing to make dietary changes or increase physical activity
* Unable to walk ¼ mile unaided without stopping
* Daily nicotine user: smoke, vape, tobacco, other
* Participants that are currently trying to lose weight via a structured weight-loss program (e.g., at a medical center, university, commercial programs)
* Participants who were a member of WW within the past 12 months
* Participants who are involved in any other research studies at this time
* Weight loss of ≥ 5 kg (11 lb) in the previous 6 months
* Reported health problems that make weight loss or unsupervised exercise unsafe or unreasonable (e.g., chronic pain, orthopedic limitations, heart problems)
* Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months
* Taking any prescription medication with known effects on appetite or weight (e.g., oral steroids, weight loss medications such as Qysmia, Contrave, Phentermine (Adipex-P, Lomaira) and others except for subjects on a stable dose of Selective serotonin reuptake inhibitors (SSRIs) for 6 months or longer
* Chronic/inflammatory gastrointestinal disorders (irritable bowel syndrome is acceptable)
* History of heart problems (e.g., angina, bypass surgery, myocardial infarction, etc.) within previous 6 months
* Diagnosis of type 1 or type 2 diabetes
* Major surgery within the previous 6 months
* Presence of implanted cardiac defibrillator or pacemaker
* History of cancer within past 5 years or current treatment for cancer
* Hospitalization for psychiatric disorders during the past 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Diet quality (Healthy Eating Index - 2015 score) | Baseline to 6-months
  Diet quality scores (HEI-2015 total score), measured with the Automated Self-Administered Dietary Assessment Tool 24-hour dietary recalls (ASA 24)

SECONDARY OUTCOMES:
Percent (%) body weight loss | Baseline to 6-months
  Weight (lb); % body weight loss defined as baseline to 6-month weight change divided by baseline weight multiplied by 100.
Achievement of 3% weight loss | Baseline to 6-months
  Proportion of participants that achieve at least 3% body weight loss at 6 months
Achievement of 5% weight loss | Baseline to 6-months
  Proportion of participants that achieve at least 5% body weight loss at 6 months
Achievement of 10% weight loss | Baseline to 6-months
  Proportion of participants that achieve at least 10% body weight loss at 6 months
Impact of weight on quality of life | Baseline to 6-months
  Measured using the Impact of Weight on Quality of Life - Lite (IWQOL).
  The IWQOL-Lite is a reliable and valid brief measure of quality of life in people with obesity. There are 31 items rated on a Likert scale 5-Always True to 1-Never True. Items are broken into subscales for physical function, self-esteem, sexual life, public distress, and work. Subscale scores and total score range from 0-100, with higher scores reflecting better levels of functioning.
Feelings of hunger over the past 7 days | Baseline to 6-months
  Measured using a Hunger Visual Analog scale (VAS) which includes a question that asks participants to rate how hungry they felt over the past week on a horizontal line with endpoints of "Not at all hungry" (0) to "Extremely hungry" (100). VAS are scored by measuring in where the participant places their tick mark on the horizontal line with endpoints of 0-100. Higher scores indicate greater feelings of hunger.
Food cravings | Baseline to 6-months
  Measured using the Food-craving Inventory (FCI-II). The FCI-II is a validated 33-item self-report measure that assesses the subjective experience of food craving across 33 different foods. The FCI-II assesses the frequency of cravings for a specified food with a five-point Likert scale (1, never; 2, rarely; 3, sometimes; 4, often; 5, always) and consists of 5 factors: high fats, sweets, carbohydrates/starches, fast food fats, & fruits and vegetables, that constitute the total food craving inventory score which averages all 33 items. Scores can range between 1 and 5, with higher scores indicating greater frequency of cravings.
Self-reported physical activity over the past 7 days | Baseline to 6-months
  Measured using the Global Physical Activity Questionnaire (GPAQ). The GPAQ collects information on physical activity participation in the following domains: activity at work, travel to- and from- places, recreational activities, and sedentary behavior. From these inputs, the minutes per week spent in moderate activity, vigorous activity, moderate and vigorous activity, and sedentary behavior can be calculated.
Self-reported Wellbeing | Baseline to 6-months
  Measured using the World Health Organization Well-being Index-5 (WHO-5). The WHO-5 consists of five statements rated by study participants with a Likert Scale: All of the time=5, Most of the time=4, More than half of the time=3, Less than half of the time=2, Some of the time=1, At no time=0. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Perceived stress | Baseline to 6-months
  Measured using the Perceived Stress Scale (PSS). The 10-item PSS measures the extent to which a participant's life is unpredictable, uncontrollable, and overloading. It was designed for use in older adolescents and adults, and is considered to have adequate internal reliability and construct validity. Each question asks about how the participant has felt or thought in the past month and uses a 5-point Likert scale (0=never, 4=very often). Scores are calculated by summing responses, creating a possible score range of 0-40, with higher scores indicating greater perceived stress.
Habit strength | Baseline to 6-months
  Measured with the Self-Reported Behavioral Automaticity Index. The self-reported behavioral automaticity index (SRBAI) captures habitual patterns of behavior. Each behavior of interest is assessed by 4 items rated on a Likert scale 1-strongly disagree to 7-strongly agree.
  Scores are calculated for each behavior by taking an average of the response values, creating a possible score range between 1 and 7. Higher scores indicate greater habit strength for the behavior being measured.
Alternate Mediterranean Diet Score (AMED) | Baseline to 6-months
  The AMED score includes seven "healthy" components: a. fruits, b. vegetables, c. fish, d. legumes, e. nuts, f. whole grains, and g. ratio of monounsaturated fat to saturated fat), and two additional components: h. red and processed meat, and i. alcohol consumption.
  Each component, except alcohol, will be categorized into quintiles (Q) and positive scores to the seven healthy components will be assigned as follows: (Q1=1, Q2=2, Q3=3, Q4=4, Q5=5). Reverse scores to red and processed meat will be assigned as follows: (Q5=1, Q4=2, Q3=3, Q2=4, Q1=5).
  For alcohol consumption (g/d), points will be assigned as follows: 5-15=5, 0-5 or 15-25=4, 0 or 25-30=3, 30-35=2, and ≥35=1 for women and 10-30=5, 0-10 or 30-40=4, 0 or 40-45=3, 45-50=2, and ≥50=1 for men.
Dietary intake | Baseline to 6-months
  Macro- and micro-nutrient intakes will be measured with the validated Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool. Participants will be asked to complete three recalls at each timepoint. Participants will be asked to complete three recalls at each timepoint.
  [Time Frame; Baseline and 6-months] Measured using the measured with the Automated Self-Administered Dietary Assessment Tool 24-hour dietary recalls (ASA 24)
Self-reported sleep quality | Baseline to 6-months
  Measured with the sleep assessment module from the validated Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool
HEI-2015 component-scores | Baseline to 6-months
  Measured with the Automated Self-Administered Dietary Assessment Tool 24-hour dietary recalls (ASA24®).

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Palacios, MD, PhD, Principal Investigator — Georgia Southern
Locations (1):
- Georgia Southern University, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data used in publications will be made available in a public repository. Data will be deidentified.
Supporting Information: Study Protocol, SAP
Time Frame: Will be made public after publications.
Access Criteria: Will be public

REFERENCES:
- [Derived] Palacios AM, Lee AM, Parker C, Watts CQ, Dickinson SL, Henschel B, Anderson G, Kersey JX, Allison DB, Foster GD, Cardel MI. Effectiveness of a digital weight management program on diet quality: a randomized controlled trial. Am J Clin Nutr. 2025 Sep;122(3):830-840. doi: 10.1016/j.ajcnut.2025.06.024. Epub 2025 Jul 1. PMID 40609748